CLINICAL TRIAL: NCT05109416
Title: Glossopharyngeal Nerve Block on Post Tonsillectomy Pain Among Egyptian Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, basem saed abdalla, Resident, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 59:4/2021
Record Dates: First submitted 2021-10-29; First posted 2021-11-05 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Post Tonsillectomy Pain
Keywords: Glossopharyngeal nerve block
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Children will receive bupivacaine 0.5% ( 1 mg / kg ) ,divided in each side , by infiltration through anterior and posterior approaches to block glossopharyngeal nerve
  Interventions: Drug: Bupivacaine Hydrochloride 0.5% Injection Solution
- Group B (Placebo Comparator): Children will receive sterile saline 0.9 , 5 cm in each side , by infiltration through anterior and posterior approaches
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride 0.5% Injection Solution — Local anesthetic
  Other Names: Marcaine
  Arms: Group A
Drug: Saline 0.9% — Isotonic crystaloid
  Other Names: Saline 0.9 %
  Arms: Group B

SUMMARY:
Tonsillectomy is one of most common performed surgical procedure in children . tonsillectomy or adenotonsillectomy have high incidence of Post operative pain , it is very important and significant problem because it can lead to decrease oral intake and dehydration

DETAILED DESCRIPTION:
Tonsillectomy is one of the most common performed surgical procedure in children. Tonsillectomy or adenotonsillectomy have high incidence of Post operative pain incidence . There is still debate about the optimal analgesia for this common procedure , different methods have been described including intraoperative anesthetic pain regimens , adjustment of surgical technique , intraoperative local anesthetic injection and use of pharmacotherapy post operative .

The main goal of the preventive analgesia is the pain releif with minimum side effect . The objective of this study is to investigate and compare the effect of Glossopharyngeal nerve block for relief of pain on children following adenotonsillectomy .

This is prospective , double blinded , randomized study

ELIGIBILITY:
Inclusion Criteria:

* average weight is 10_50 kg
* patient is generally stable
* indication of tonsillectomy is recurrent tonsillitis
* Ability to self report pain

Exclusion Criteria:

* Hypersensitivity to bupivacaine
* Obstructive sleep apnea syndrome
* Pulmonary or cardic diseases

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2021-10-17 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
The first call for analgesia | In 24 hours
  Pain assessment using VAS scale

SECONDARY OUTCOMES:
The analgesic consumption | In 24 hours
  The total analgesic consumption for pain rest and swallowing

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medcine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No